CLINICAL TRIAL: NCT01203462
Title: A Probiotic Double-blind Randomized Placebo Crossover Trial of Colonic Transit Time in Adult Females, The PRIDE Study The Study to Determine the Effects of Probiotics on Regulation and Improving Digestive hEalth
Brief Title: The PRIDE Study Probiotics on Regulation and Improving Digestive hEalth
Acronym: PRIDE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Cargill (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2010-402
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2012-12

CONDITIONS: Digestive Irregularity; Digestive Discomfort; History of Straining During Bowel Movements; History of Hard or Lumpy Stools

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bifidobacterium supplemented yogurt (Experimental): Bifidobacterium supplemented (minimum dosage of 1E+10cfu/serving) vanilla flavored yogurt containing starter cultures: Streptococcus thermophilus and Lactobacillus delbrueckii subsp. Bulgaricus
  Interventions: Other: Probiotic strain of Bifidobacterium
- Placebo Yogurt (Placebo Comparator): Vanilla flavored yogurt containing starter cultures Streptococcus thermophilus and Lactobacillus delbrueckii subsp. Bulgaricus
  Interventions: Other: No Bifidobacterium

INTERVENTIONS:
Other: Probiotic strain of Bifidobacterium — 4 ounces (113g) of yogurt per day, for 14 days. Minimum Bifidobacterium dose of 1E+10 cfu/serving.
  Arms: Bifidobacterium supplemented yogurt
Other: No Bifidobacterium — 4 ounces (113g) of yogurt per day, for 14 days. No bifidobacterium added.
  Arms: Placebo Yogurt

SUMMARY:
The purpose of this study is to determine the effect of probiotic supplemented yogurt in reducing colonic transit time (CTT) in females between the ages of 18-65 years old. Two yogurts will be administered, one containing a specific strain of probiotic in the Bifidobacterium genus and the other without the probiotic supplement. It is hypothesized that subjects receiving the probiotic supplemented yogurt will experience reduced CTT and improved gastrointestinal comfort and quality of life compared to those receiving the non-probiotic supplemented yogurt.

ELIGIBILITY:
Inclusion Criteria:

* Being female
* Ability to speak and write English or Spanish
* Willingness to refrain from specified probiotic supplements, during the 12 week trial (a list of prohibited products will be provided)
* Have access to refrigeration and phone
* Have a history of straining during bowel movements
* Have a history of lumpy or hard stools

Exclusion Criteria:

* Presence of an allergy or intolerance to any ingredients in yogurt
* Morbid obesity, defined as a BMI>40
* Having inflammatory bowel disease
* Having a history of malabsorption syndrome
* Immunodeficiency, such as HIV or currently receiving chemotherapy
* Consumption of any medications used to treat, prevent or cure diarrhea in the last month
* Consumption of any medications used to treat, prevent or cure constipation in the last month
* Diabetes mellitus
* Thyroid disorders, including hypo- or hyperthyroidism
* History of gastric, small bowel or colonic resection
* Documented history of gastric emptying disorder
* Consumption of narcotics, antipsychotic medications, or verapamil in the last month
* Known pelvic outlet obstruction
* Antibiotic usage within 4 weeks of enrollment
* Pregnancy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2010-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Colonic Transit Time | 90 days

SECONDARY OUTCOMES:
Frequency of bowel movements (daily) | 90 days
Stool consistency (daily) | 90 days
Well being as assessed by agreed upon quality of life instrument | 90 days
Dietary intake survey | 90 days
Tolerance | 90 days
  by questionnaire: e.g. bloating
Rome criteria | 90 days
Bristol criteria | 90 days
Recovery of the probiotic in the faeces (quantitative measure) | 90 days
Bacterial composition of the fecal flora | 90 days
Adverse events | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Dan Merenstein, MD, Principal Investigator — Georgetown University; Caren Palese, MD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University Department of Family Medicine, Research Division, Washington D.C., District of Columbia, United States